CLINICAL TRIAL: NCT05583981
Title: Stakeholder Assessment of Implementing the Commission on Cancer Operative Standards for Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ko Un Park, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-21198; NCI-2021-08725 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1K08CA263488-01A1 (NIH); 202010121 (Other Grant/Funding Number: Alliance NCTN Foundation)
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (interview): Participants participate in interview over 30-60 minutes.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Participate in interview

SUMMARY:
This study investigates the barriers to implementing breast Synoptic Operative Reports. Information from this study may help researchers identify performance objectives for the breast Synoptic Operative Reports to be adopted, implemented and continued.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify and describe barriers to implementing breast Synoptic Operative Reports (SOR) from multiple constructs.

Ia. Identify performance objectives - who must do what - for the breast SOR to be adopted, implemented, and continued.

OUTLINE:

Participants participate in interview over 30-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 18 years
* Available phone or device for contact
* English speaking
* Works at Commission on Cancer (CoC) - accredited cancer program

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Key stakeholders (e.g. electronic medical record [EMR] engineer, Cancer Liaison Physician [CLP], breast surgeon, and cancer registrar administrator) from Ohio State University and 3 other Commission on Cancer (CoC)-accredited cancer programs
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Barriers to implementing breast Synoptic Operative Reports | Up to 2 years
  This is a qualitative study in which we will conduct in-depth, semi-structured interviews with key stakeholders. A template analysis identifying priori themes will be used, then coding for impact and/or implementation strategy.
Performance objectives for the breast Synoptic Operative Reports to be adopted, implemented, and continued | Up to 2 years
  This is a qualitative study in which we will conduct in-depth, semi-structured interviews with key stakeholders.A template analysis identifying priori themes will be used, then coding for impact and/or implementation strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Ko Un Park, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT05583981/ICF_000.pdf